CLINICAL TRIAL: NCT00003311
Title: Phase II CCOP Trial of High Dose Methotrexate/ARA-C and HCVAD for Newly Diagnosed Nodular and Diffuse Mantle Cell Lymphoma and Their Blastic Variants
Brief Title: Combination Chemotherapy in Treating Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066258; MDA-DM-97200; NCI-T97-0101; DM97-200 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2003-04-25 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (Experimental): Methotrexate IV over 24 hours on day 1. Cytarabine is administered IV over 2 hours every 12 hours on days 2 and 3. Filgrastim (G-CSF) is administered subcutaneously (SC) daily beginning on day 4 and continuing until blood counts recover. Treatment repeats every 21 days for up to 8 courses.
  Interventions: Biological: filgrastim; Drug: cytarabine; Drug: methotrexate
- Regimen B (Experimental): Cyclophosphamide IV over 3 hours every 12 hours on days 1-3. Doxorubicin is administered IV over 24 hours on days 4 and 5. Vincristine is administered IV over 30 minutes on days 4 and 11. Dexamethasone is administered orally or IV on days 1-4 and 11-14. G-CSF is administered SC beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for up to 7 courses.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
  Arms: Regimen B
Drug: cytarabine
  Arms: Regimen A
Drug: dexamethasone
  Arms: Regimen B
Drug: doxorubicin hydrochloride
  Arms: Regimen B
Drug: methotrexate
  Arms: Regimen A
Drug: vincristine sulfate
  Arms: Regimen B

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of different regimens of combination chemotherapy in treating patients with newly diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the complete response rate and duration of response in patients with newly diagnosed diffuse or nodular mantle cell lymphoma or their blastic variant treated with high-dose methotrexate and cytarabine and high-dose cyclophosphamide, dexamethasone, doxorubicin, and vincristine (HCVAD).

OUTLINE: This is a multicenter study. Patients may receive either regimen A or both regimen A and regimen B, depending upon response.

* Regimen A: Patients receive methotrexate IV over 24 hours on day 1. Cytarabine is administered IV over 2 hours every 12 hours on days 2 and 3. Filgrastim (G-CSF) is administered subcutaneously (SC) daily beginning on day 4 and continuing until blood counts recover. Treatment repeats every 21 days for up to 8 courses.
* Regimen B: Patients receive cyclophosphamide IV over 3 hours every 12 hours on days 1-3. Doxorubicin is administered IV over 24 hours on days 4 and 5. Vincristine is administered IV over 30 minutes on days 4 and 11. Dexamethasone is administered orally or IV on days 1-4 and 11-14. G-CSF is administered SC beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for up to 7 courses.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 21-45 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously untreated nodular or diffuse mantle cell lymphoma or their blastic variant
* No CNS involvement
* Not a candidate for stem cell transplantation or refuses one

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3*
* Platelet count greater than 100,000/mm^3* NOTE: * Unless lymphoma involvement

Hepatic:

* Bilirubin less than 1.5 mg/dL (unless lymphoma involvement)

Renal:

* Creatinine less than 2.0 mg/dL (unless lymphoma involvement)

Cardiovascular:

* Cardiac ejection fraction at least 50% (for patients over age 40)

Other:

* Must be willing to receive blood transfusion
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other co-morbid medical or psychiatric illness that would preclude treatment
* No prior or concurrent malignancy with poor prognosis (less than 90% probability of survival at 5 years)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1998-05-20 (Actual); Primary Completion 2007-04-18 (Actual); Study Completion 2007-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Romaguera, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States